CLINICAL TRIAL: NCT03431272
Title: Use of 5.0% Lifitegrast Ophthalmic Solution for the Treatment of Dry Eye Disease in Contact Lens Wearers
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: no longer interest / resources to start study
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Shire (Industry)
Responsible Party: Principal Investigator, Jason Nichols, Principal Investigator, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F49384759
Record Dates: First submitted 2018-02-06; First posted 2018-02-13 (Actual); Last update posted 2018-10-25 (Actual); Status verified 2018-10

CONDITIONS: Contact Lens Dry Eye
Keywords: contact lens, discomfort, dry eye
MeSH Terms: conditions — Dry Eye Syndromes | interventions — lifitegrast

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (Experimental): lifitegrast ophthalmic solution 5.0%, to be instilled 1 drop in each eye, twice a day
  Interventions: Drug: Lifitegrast

INTERVENTIONS:
Drug: Lifitegrast — Eye drop
  Other Names: Xiidra

SUMMARY:
Discomfort with contact lens wear is the biggest reason why people stop wearing contact lenses. The investigators believe that inflammation is one of the causes of discomfort, and by blocking the inflammation using lifitegrast, the investigators may be able to relieve some of that discomfort. This study will enroll 50 subjects with contact lens discomfort and will receive lifitegrast to use over a period of approximately 3 months.

DETAILED DESCRIPTION:
The most common reason for contact lens drop out is ocular discomfort, with patients identifying dryness as the major reason. Currently, many patients with contact lens dry eye (CLDE) utilize rewetting drops to relieve their symptoms. The problem with rewetting drops is that they fail as they are transient, and do not address the inflammatory component of contact lens discomfort. Lifitegrast 5.0% ophthalmic solution was approved and is now marketed as Xiidra, for the treatment of signs and symptoms of dry eye disease. Lifitegrast works by reducing inflammation, which suggests that it may be effective in patients with contact lens dry eye. More specifically, lifitegrast may work by blocking the interaction between ICAM-1 and LFA-1, which leads to a decrease in the activation and recruitment of T-cells, and a decrease in pro-inflammatory cytokines.

The safety and efficacy of Xiidra has been studied in four, 12 week clinical trials involving over 2,100 patients. Each study assessed the effects of Xiidra on symptoms using an Eye Dryness Score (EDS), which is a visual analogue ranging from 0 (no discomfort) to 100 (maximal discomfort). In two of those studies, lifitegrast was shown to improve symptom relief at weeks 2, 6, and 12 compared to the placebo (https://www.xiidra-ecp.com/efficacy-symptom-improvement).

Each of the four clinical trials mentioned above also assessed clinical signs of dry eye disease, with a particular focus on inferior corneal staining graded on 0.5 unit increments on a 0 (no staining) to 4 scale (coalescent). In three of the four clinical trials, lifitegrast reduced inferior corneal staining by week 12, compared to placebo (https://www.xiidra-ecp.com/efficacy-treating-signs).

Contact lens dry eye is mediated by significant symptoms of ocular surface dryness, in addition to similar clinical signs of dry eye disease such as corneal staining and inflammation. Thus, the purpose of this interventional study is to examine the effect of lifitegrast ophthalmic solution in subjects with contact lens dry eye.

ELIGIBILITY:
Inclusion Criteria:

* Has provided informed consent.
* Age ≥ 18 years.
* Have a diagnosis of CLDE based on Contact Lens Dry Eye Questionnaire (CLDEQ) results:

Answer to question #10 of "Yes" and score >-0.13, or Answer to Question #10 of "No" and score > 1.27, or Answer to #10 of "Unsure" and score > 1.44

* Have a score of ≥ 2 on the Ocular Dryness Assessment at Visit 1.
* Are willing and able to follow instructions and can be present for the required study visits for the duration of the study.
* Are willing to avoid restricted medications for the time frames indicated during the study.
* Wears soft contact lenses at least 4 days a week for at least 5 hours per day using the same brand of contact lenses for at least the last 30 days.

Exclusion Criteria:

* Have a history of significant adverse reaction to lifitegrast or other components of the drug product, or contraindication to the use of lifitegrast or other components of the drug product.
* Have changed the brand or material or design of soft contact lenses or care solutions within 30 days prior to screening or anticipates the need to change current type/brand of contact lenses or care solutions throughout the 84-day study.
* Use contact lenses overnight.
* Use rigid gas permeable contact lenses or hybrid lenses.
* Have any uncontrolled systemic diseases that in the investigator's opinion could be expected to interfere with the study.
* Have had cauterization of the punctum or have had punctal plugs (silicone or collagen) inserted or removed within the 90 days prior to the screening.
* Have any active ongoing ocular infection, ocular disease or condition that would require treatment with topical ophthalmic medications.
* Require any topically delivered ophthalmic medication for any condition during the study. This includes any preserved or unpreserved rewetting drops or artificial tears. The subject must not have used ophthalmic prescription medications for at least 30 continuous days prior to Visit 1, and must not have used rewetting drops or artificial tears for at least 5 continuous days prior to Visit 1.
* Have recently started taking omega-3 fatty acids supplements within the past 2 months.
* Are taking Omega-3 fatty acids supplements but unable to maintain consistent dosage for the duration of the study.
* Are unwilling or unable to comply with the protocol.
* Have been exposed to any investigational drug within the preceding 30 days.
* Are an employee of the site that is directly involved in the management, administration, or support of this study or be an immediate family member of the same.
* If female, participant must be non-pregnant and non-lactating, and those of childbearing potential must be using an acceptable method of birth control (i.e. an Intrauterine Contraceptive Device with failure rate of <1%, hormonal contraceptives, or a barrier method.) If a female subject is abstinent, she must agree to use one of the acceptable contraceptive methods if she becomes sexually active.
* Have a clinically significant ophthalmic abnormality, infection, or disease noted by subject history or examination that would otherwise contraindicate contact lens wear and/or the use of lifitegrast (i.e., ≤ grade 3 giant papillary conjunctivitis, active ocular allergies, conjunctivitis, keratitis, uveitis).
* Have had a history of corneal surgery (corneal transplants, LASIK, PRK).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-11-01 (Estimated); Primary Completion 2018-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of hours related to comfort in wearing contact lenses. | Baseline to Week 12.
  The amount of comfortable lens wear time averaged over the 12th week of lens wear as reported with participant diary.

SECONDARY OUTCOMES:
Number of hours related to comfort in wearing contact lenses. | Baseline to Week 2.
  The amount of comfortable lens wear time averaged over the 2nd week of lens wear as reported with participant diary.
Number of hours related to comfort in wearing contact lenses. | Baseline to Week 6.
  The amount of comfortable lens wear time averaged over the 6th week of lens wear as reported with participant diary.
Number of hours related to total contact lens wear. | Baseline to Week 2.
  The amount of total lens wear time averaged over the 2nd week of lens wear as reported with participant diary.
Number of hours related to total contact lens wear. | Baseline to Week 6.
  The amount of total lens wear time averaged over the 6th week of lens wear as reported with participant diary.
Number of hours related to total contact lens wear | Baseline to Week 12
  The amount of total lens wear time averaged over the 12th week of lens wear as reported with participant diary.
Number of hours of overall eye dryness in the morning. | Baseline to Week 2.
  The amount of overall eye dryness experienced in the morning, averaged over the 2nd week of lens wear as reported with participant diary.
Number of hours of overall eye dryness in the morning. | Baseline to Week 6th.
  The amount of overall eye dryness experienced in the morning, averaged over the 6th week of lens wear as reported with participant diary.
Number of hours of overall eye dryness in the morning. | Baseline to Week 12th.
  The amount of overall eye dryness experienced in the morning, averaged over the 12th week of lens wear as reported with participant diary.
Number of hours of overall eye dryness in the evening. | Baseline to Week 2.
  The amount of overall eye dryness experienced in the evening, averaged over the 2nd week of lens wear as reported with participant diary.
Number of hours of overall eye dryness in the evening | Baseline to Week 6
  The amount of overall eye dryness experienced in the evening, averaged over the 6th week of lens wear as reported with participant diary
Number of hours of overall eye dryness in the evening. | Baseline to Week 12.
  The amount of overall eye dryness experienced in the evening, averaged over the 12th week of lens wear as reported with participant diary.
Change in Contact Lens Dry Eye diagnosis. | Baseline to Week 2.
  The participant diagnosis is made using the Contact Lens Dry Eye Questionnaire at Week 2.
Change in Contact Lens Dry Eye diagnosis. | Baseline to Week 6.
  The participant diagnosis is made using the Contact Lens Dry Eye Questionnaire at Week 6.
Change in Contact Lens Dry Eye diagnosis. | Baseline to Week 12.
  The participant diagnosis is made using the Contact Lens Dry Eye Questionnaire at Week 12.

CONTACTS AND LOCATIONS:
Overall Officials: Jason J Nichols, OD PhD MPH, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Richdale K, Sinnott LT, Skadahl E, Nichols JJ. Frequency of and factors associated with contact lens dissatisfaction and discontinuation. Cornea. 2007 Feb;26(2):168-74. doi: 10.1097/01.ico.0000248382.32143.86. PMID 17251807
- [Background] Efron N. Contact lens wear is intrinsically inflammatory. Clin Exp Optom. 2017 Jan;100(1):3-19. doi: 10.1111/cxo.12487. Epub 2016 Nov 2. PMID 27806431
- [Background] Gao J, Morgan G, Tieu D, Schwalb TA, Luo JY, Wheeler LA, Stern ME. ICAM-1 expression predisposes ocular tissues to immune-based inflammation in dry eye patients and Sjogrens syndrome-like MRL/lpr mice. Exp Eye Res. 2004 Apr;78(4):823-35. doi: 10.1016/j.exer.2003.10.024. PMID 15037117
- [Background] Zhang Y, Wang H. Integrin signalling and function in immune cells. Immunology. 2012 Apr;135(4):268-75. doi: 10.1111/j.1365-2567.2011.03549.x. PMID 22211918
- [Background] Shire. Efficacy Info. 2017; https://www.xiidra-ecp.com/efficacy-symptom-improvement. Accessed 12/21/2017, 2017.
- [Background] Shire. Xiidra and ICSS. 2017; https://www.xiidra-ecp.com/efficacy-treating-signs. Accessed 12/21/2017, 2017.
- [Background] Shire. Mechanism of Action. 2017; https://www.xiidra-ecp.com/mechanism-of-action. Accessed 12/21/2017, 2017.
- [Background] U.S. Food & Drug Administration. What is a Serious Adverse Event? 2016; https://www.fda.gov/Safety/MedWatch/HowToReport/ucm053087.htm. Accessed 12/11/2017, 2017.